CLINICAL TRIAL: NCT07126548
Title: A Pragmatic Clinical Trial to Evaluate the Effect of a Point of Prostate Cancer Diagnosis (PPCD) Virtual Reality Assistant (ViRA) in Supporting Newly Diagnosed Black Men
Brief Title: A Point of Prostate Cancer Diagnosis Virtual Reality Assistant Intervention in Supporting Newly Diagnosed Black Men
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MC250501; NCI-2025-04864 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-013879 (Other: Mayo Clinic Institutional Review Board); MC250501 (Other: Mayo Clinic); HT94252411104 (Other Grant/Funding Number: Department of Defense); PC230672P11 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Masking Description: Protocol indicated this being a two-arm randomized, single-blind clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (delayed-start intervention [ViRA application]) (Experimental): Patients receive standard care and then receive access to the ViRA app (on a VR headset, smartphone, iPAD or computer) and are presented with short screening questions, which an AI engine uses to recommend personalized and culturally tailored VR ready CaP interventions facilitated by a digital human character (CaP survivor, physician, or a psycho-oncologist) 3 months later on study.
  Interventions: Other: Best Practice; Other: Discussion; Other: Survey Administration; Procedure: Virtual Reality
- Arm II (ViRA application) (Experimental): Patients receive access to the ViRA app (on a VR headset, smartphone, iPAD or computer) and are presented with short screening questions, which an AI engine uses to recommend personalized and culturally tailored VR ready CaP interventions facilitated by a digital human character (CaP survivor, physician, or a psycho-oncologist) on study.
  Interventions: Other: Discussion; Other: Survey Administration; Procedure: Virtual Reality

INTERVENTIONS:
Other: Best Practice — Receive standard care
  Other Names: standard of care; standard therapy
  Arms: Arm I (delayed-start intervention [ViRA application])
Other: Discussion — Ancillary studies
  Other Names: Discuss
Other: Survey Administration — Ancillary studies
Procedure: Virtual Reality — Receive access to ViRA application
  Other Names: VR

SUMMARY:
This clinical trial tests how well a point of prostate cancer diagnosis (PPCD) virtual reality assistant (ViRA) intervention works in supporting Black men with newly diagnosed prostate cancer. Cancer is the second leading cause of death for African American/Black men, with prostate cancer leading in estimated new cancer cases and second in estimated new cancer deaths. Over 40,000 African American/Black men are diagnosed with prostate cancer annually, with 1 in 6 lifetime probability of developing prostate cancer compared to 1 in 8 probability in White men. The PPCD ViRA provides psycho-oncology support, social determinants of health navigation and emotional support for ethnically diverse African American/Black men newly diagnosed with prostate cancer using artificial intelligence and augmented reality. Using PPCD ViRA may close the prostate cancer care gap for African American/Black men across the cancer continuum and provide emotional, educational, and resource needs of this population when they are visiting a doctor about their prostate health or prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the effectiveness of the PPCD ViRA (i) on the delivery of PPCD support in a clinic setting, at home and community setting; and (ii) in providing social determinants of health (SDOH) navigation, emotional support and psycho-oncology support for African American/Black men (AA/BM) newly diagnosed with prostate cancer (CaP).

II. Assess the effectiveness of the PPCD ViRA in reducing emotional distress and improving other patient reported outcomes (PROs).

III. Using a mixed-method approach, explore the factors that uniquely influence the implementation of the PPCD ViRA in a clinic setting, at home and community setting.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (DELAYED-START INTERVENTION): Patients receive standard care and then receive access to the ViRA application (app) (on a [virtual reality] VR headset, smartphone, iPAD or computer) and are presented with short screening questions, which an AI engine uses to recommend personalized and culturally tailored VR ready CaP interventions facilitated by a digital human character (CaP survivor, physician, or a psycho-oncologist) 3 months later on study.

ARM II (EARLY START INTERVENTION): Patients receive access to the ViRA app (on a VR headset, smartphone, iPAD or computer) and are presented with short screening questions, which an AI engine uses to recommend personalized and culturally tailored VR ready CaP interventions facilitated by a digital human character (CaP survivor, physician, or a psycho-oncologist) on study.

After completion of study intervention, patients are followed up at 1, 3, 6, 9 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* African American/Black male
* Diagnosed with CaP within two months
* Be a patient at a participating clinic or affiliates with one of our community sites
* Consent to participating in the study

Exclusion Criteria:

* Do not speak or understand English
* Unable to read or write

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-09-02 (Estimated); Study Completion 2029-09-02 (Estimated)

PRIMARY OUTCOMES:
Reach - enrollment | Baseline
  Reach of the point of prostate cancer diagnosis (PPCD) virtual reality assistant (ViRA) will be measured by the number of AA/BM who enroll in the study when offered.
Reach - acceptance of ViRA | Baseline
  Reach of the PPCD ViRA will be measured by the % of AA/BM who accept the ViRA when offered.
Reach - initiation of ViRA | Baseline, 1 month, 3 months, 6 months, 9 months, 12 months
  Reach of the PPCD ViRA will be measured by the number of AA/BM who initiate the ViRA at the clinic vs. home vs. community setting.
Utilization of the PPCD ViRA | Baseline, 1 month, 3 months, 6 months, 9 months, 12 months
  Will be measured by total # of AA/BM who used the Vira at least once a week.

SECONDARY OUTCOMES:
Change in social determinants of health (SDOH) navigation | Baseline, 1 month, 3 months, 6 months, 9 months, 12 months
  Will be assessed by participant self-reported ability to find help for daily needs such as food, housing, reliable transportation for medical appointments.
Change in emotional support | Baseline, 1 month, 3 months, 6 months, 9 months, 12 months
  Will be measured using the Positive Affect and Negative Affect Schedule-Expanded Form (PANAS-X), a 60-item questionnaire designed to measure a person's emotional state, both positive and negative, during a specific time frame. Participants rate how they feel on a 5-point Likert scale for each item (e.g., "right now" or "in general"). For the total positive score, a higher score indicates more of a positive affect. For the total negative score, a lower score indicates less of a negative affect.
Psycho-oncology support | Baseline, 1 month, 3 months, 6 months, 9 months, 12 months
  Assessed by providers using National Comprehensive Cancer Network (NCCN) Guidelines Version 1.2024 Distress Management.

CONTACTS AND LOCATIONS:
Overall Officials: Folakemi T. Odedina, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials